CLINICAL TRIAL: NCT04872686
Title: A Multicenter, Single Blind, Randomized Controlled Trial of Virucidal Effect of Polyvinyl Pyrrol-Iodine on SARS-CoV-2 as Well as Safety of Its Application on Nasopharynx & Oropharynx of COVID-19 Positive Patients
Brief Title: Virucidal Effect of PVP-I on COVID-19 and as Well as Safety of Its Application on Nasopharynx & Oropharynx
Acronym: COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DR. MALA KHAN (Other Government)
Collaborators: Bangladesh Reference Institute of Chemical Measurements (BRICM) (Other Government)
Responsible Party: Sponsor-Investigator, DR. MALA KHAN, Director General and Chief ScientificOfficer, Bangladesh Reference Institute of Chemical Measurements (BRICM)
Organization: Bangladesh Reference Institute of Chemical Measurements (BRICM) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BRiCM LABS BANGASAFE SPRAY
Record Dates: First submitted 2021-04-26; First posted 2021-05-04 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Virus Infection, RNA; Effect of Drug; Efficacy, Self
Keywords: Viral load; PVP-I; SARS-CoV-2; Shelf-life; Stability
MeSH Terms: conditions — RNA Virus Infections | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Oral and nasal spray to moderately ill COVID-19 positive patient (Experimental): Drug Name: Povidone-Iodine Dosage form: 0.6% Povidone-Iodine Dosage: 2 puff 0.6% PVP-I in each nostril and 2 puff inside mouth Frequency and duration: Single
  Interventions: Drug: 0.6% PVP-I oral and nasal spray to moderately ill COVID-19 positive patient
- Oral and nasal spray to asymptomatic to mild COVID-19 patient having multiple comorbidity (Experimental): Drug Name: Povidone-Iodine Dosage form: 0.6% Povidone-Iodine Dosage: 2 puff 0.6% PVP-I in each nostril and 2 puff inside mouth Frequency and duration: hourly for 4 hours in a single day
  Interventions: Drug: 0.6% PVP-I Oral and nasal spray to asymptomatic to mild COVID-19 patient having multiple comorbidity
- Oral and nasal spray to healthy volunteer (Experimental): Drug Name: Povidone-Iodine Dosage form: 0.6% Povidone-Iodine Dosage: 2 puff 0.6% PVP-I in each nostril and 2 puff inside mouth Frequency and duration: 3-4 times interval but not more than 4 times a day for 30 days
  Interventions: Drug: 0.6% PVP-I Oral and nasal spray to healthy volunteer
- Oral and nasal spray by distilled water to control group (Placebo Comparator): Placebo comparator: Distilled water Dosage form: Oral and Nasal spray will be provided by Distilled water
  Interventions: Other: Oral and nasal spray by distilled water to control group

INTERVENTIONS:
Drug: 0.6% PVP-I oral and nasal spray to moderately ill COVID-19 positive patient — Number of participants 768 COVID-19 positive, moderately ill admitted patient who will receive intervention
  Step 1: Enrollment of the study populations by applying inclusion and exclusion criteria Step 2: Randomization to allocate experimental and controlled group by using table of random number Step 3: Application of 0.6% PVP-I spray to experimental group and distilled water to control group Step 4: Follow up (waiting for 2-5 minutes) Step 5: Collection of nasopharyngeal and oropharyngealsawab for RT-PCR test for both group Step 6: Observation of the patients for 30 minutes for possible early adverse effects (if any) and subsequent management (if needed).
  Step 7: Analysis data collection, data processing and analysis by using SPSS software.
  Other Names: Group A
  Arms: Oral and nasal spray to moderately ill COVID-19 positive patient
Drug: 0.6% PVP-I Oral and nasal spray to asymptomatic to mild COVID-19 patient having multiple comorbidity — Number of participants 20 asymptomatic to mild COVID -19 patients having multiple comorbidity who will receive intervention
  Step 1: Selection of 20 patients randomly with no or mild symptoms and obtain their consent for the further tests.
  Step 2: Collection of 2nd, 3rd and 4th sample from nasopharynx and oropharynx hourly Step 3: Data collection, data processing and analysis by using SPSS software
  Other Names: Group B
  Arms: Oral and nasal spray to asymptomatic to mild COVID-19 patient having multiple comorbidity
Drug: 0.6% PVP-I Oral and nasal spray to healthy volunteer — Number of participants 10 healthy individual who accept intervention 0.6% PVP-I oronasal spray
  Step 1: Selection of 10 healthy volunteers randomly who will be selected for using 0.6% PVP-I Oro-Nasal spray 2 puff inside both nostrils and mouth 3 to 4 times a day for one month.
  Step 2: Collection of blood & urine of participants on day 0, 10, 20, 30 for determination of any change in biochemical marker (thyroid, kidney and liver functions will be done) Step 3: Data collection, data processing and analysis by using SPSS software
  Other Names: Group C
  Arms: Oral and nasal spray to healthy volunteer
Other: Oral and nasal spray by distilled water to control group — Placebo comparator: Distilled Water Oral and Nasal spray will be provided by Distilled water to control group
  Other Names: Control Group
  Arms: Oral and nasal spray by distilled water to control group

SUMMARY:
The COVID-19 pandemic is the defining global health crisis of our time and the greatest challenge we have faced since World War-II.Corona virus is transmitted via respiratory droplets or aerosol, produced from sneezing or coughing of infected persons to healthy individual through mouth, nose and eye. PVP-I gargle/spray used in throat and nose are shown to have broad spectrum antimicrobial activity and may have preventive effect on SARS-CoV-2.

0.6% PVP-I oro-nasal spray phase 3 clinical trial will be conducted in three dedicated Covid-19 hospitals namely Dhaka Medical College Hospital, Kurmitola General Hospital, Kuwait-Moitree Hospital. Chemical compound of the oro-nasal spray which was developed and tested at Bangladesh Reference Institute for Chemical Measurements, for its quality control/ quality assurance, shelf life and related stability following GLP guideline.

This study aims to evaluate virucidal efficacy of 0.6% PVP-I against SARS-CoV-2 along with its safe uses in oronasal mucosa of healthy and SARS-CoV-2 exposed persons.

The participant will be divided into three groups: Group A 768 COVID-19 positive, moderately ill admitted patient who will receive intervention once. Group B 20 asymptomatic to mild COVID-19 patients having multiple comorbidity will receive intervention 4 times hourly and Group C 10 healthy individual who accept intervention 0.6% PVP-I oronasal spray 3-4 times interval in a day for 30 days. Placebo will be used among control group for better comparison.

The chemical which will be used in this study is available inside the country and also registered to open use in Bangladesh. BRiCM ensures raw material & impurities characterization as per BP 2019, AOAC and AWWA and determination of shelf life by performing the stability studies will be conducted according to Stability Zone Iva and ICH guidelines.

A written consent will be taken by concern participant and a short interview will be taken on the spot prior to intervention. Participant's medical documents will be used and swab from nasopharynx & oropharynx will be taken for performing necessary test (RT-PCR) to confirm viral presence.

There is no potential risk for application of this oro-nasal spray. Even though if any adverse reaction occur while using the oro-nasal spray, necessary medical management will be carried out in the respected hospital.

DETAILED DESCRIPTION:
Introduction:

COVID-19 pandemic is the defining global health crisis of our time and the greatest challenge we have faced since World War Two. We have now reached the tragic milestone of two million deaths, and the human family is suffering under an almost intolerable burden of loss.

Background Information:

1. Description of Bangasafe (proposed name) Oro-Nasal Spray: The spray contains PVP-I is a water-soluble iodophor that consists of a complex between iodine and a solubilizing polymer carrier, polyvinylpyrrolidone. In aqueous solution, a dynamic equilibrium occurs between free iodine, the active virucidal agent, and the PVP-I-complex.
2. Composition: Oro-Nasal spray contains 0.6% PVP-I as an Active Pharmaceutical Ingredients (API) in sterile de-ionized water.
3. Product Development, Quality Control and Quality Assurance: Following aspects of raw materials including API, manufacturing in-process steps, finished product are to be real time monitored and produced in Bangladesh Reference Institute for Chemical Measurements,

   * Raw materials characterization: Appearance, solubility, identification, nitrogen content, iodide value, loss on drying, pH, sulphated ash and available iodine.
   * Solvent/diluent characterization: pH, conductivity, total organic carbon, heavy metal (Pb, As), endotoxin, microbial count.
   * Quality testing in several stages during product development: pH, available iodine, iodide, UV absorbance, potency.
   * Impurity profile testing: 1-Vinyl-2-pyrrolidinone, 2-Pyrrolidinone, heavy metal (Pb)
   * Accelerated & real time stability study and shelf-life determination: pH, available iodine, iodide, UV absorbance Up to 3 (three) month at 25C, 30C and 35C
4. Mode of Action: PVP itself has no microbicidal activity but rather delivers the free iodine to target cell membranes. The basic mechanism leads to strong microbicidal activity expressed by multiple modes of action as oxidation of amino acids and nucleic acids that disrupt the microbial metabolic pathways, as well as destabilization of the structural components of cell membranes, causing irreversible damage to the pathogen.
5. Dosage and Administration: Mouth & Nostril: 2 puffs, in 3-4 hours interval not more than 4 times a day.
6. How Supplied: Oro-nasal spray aqueous solution containing 0.6%PVP-I is supplied in 30ml amber color High Density Poly Ethylene (HDPE) bottle designed for pharmaceutical packaging to provide adequate protection against sun light.

Objectives of the study

1. Primary Objective

   To assess the virucidal efficacy of 0.6% PVP-I against SARS-CoV-2 in nasopharynx and oropharynx in order to use:
   * To prevent viral infection before exposure while visiting and treating COVID-19 patients, attending public gatherings, using public transport etc.
   * To prevent viral infection after exposure to COVID-19 patients
   * To reduce viral load in nasopharynx and oropharynx of COVID-19 patients which is supposed to reduce viral transmission through respiratory route
2. Secondary Objectives

   * To assess the viral load in the nasopharynx and oropharynx before and after application of 0.6% PVP-I of participants of this study.
   * To assess the duration of effectivity of 0.6% PVP-I on mucosal surface of participating COVID-19 patients by testing consecutive sample hourly upto 4hr .
   * To estimate the shelf-life and stability of 0.6 % PVP-Ioronasal spray.
   * To characterize raw materials and impurities for product development and quality control/ assurance
   * To measure the safety level of 0.6% PVP-Ioronasal sprayby biochemical analysis of participants blood & urine This study aims to evaluate virucidal efficacy of 0.6% PVP-I against SARS-CoV-2 amongst humans and its safety that is expected to contribute to save lives during this COVID-19 pandemic.

Methodology Study design It will be a Multicentre, Single blind, Randomized Controlled Trial.The participant will be divided into three groups namely Group A : 768 (384 intervention group and 384 control group) COVID-19 positive, moderately ill admitted patient will receive intervention once (2 puff 0.6% PVP-I in each nostril and mouth).

Step 1: Enrollment of the study populations by applying inclusion and exclusion criteria Step 2: Randomization to allocate experimental and controlled group by using table of random number Step 3: Application of 0.6% PVP-I spray to experimental group and distilled water to control group Step 4: Follow up (waiting for 2-5 minutes) Step 5: Collection of nasopharyngeal and oropharyngealsawab for RT-PCR test for both group Step 6: Observation of the patients for 30 minutes for possible early adverse effects (if any) and subsequent management (if needed).

Step 7: Data collection, processing and analysis by SPSS software.

Group B : 20 asymptomatic to mild Covid -19 patients having multiple comorbidity will receive intervention 4 times (2 puff 0.6% PVP-I containing oronasal spray in to each nostril and mouth).

Step 1: Selection of 20 patients randomly with no or mild symptoms and obtain their consent for the further tests.

Step 2: Collection of 2nd, 3rd and 4th sample from nasopharynx and oropharynx hourly Step 3: Data collection, processing and analysis by SPSS software

Group C : 10 healthy individual who accept intervention 0.6% PVP-I oronasal spray 3-4 times interval but not more than 4 time a day for 30 days.

Step 1: Selection of 10 healthy volunteers randomly for using 0.6% PVP-I Oro-Nasal spray 2 puff inside both nostrils and mouth 3 to 4 times a day for one month.

Step 2: Collection of blood & urine of participants on day 0, 10, 20, 30 for determination of any change in biochemical marker (thyroid, kidney and liver functions will be done) Step 3: Data collection, processing and analysis by SPSS software

Raw material & impurities characterization

* PVP-I collection from approved vendor with certificate of analysis (CoA)
* Characterization tests of PVP-I such as appearance, identification, solubility, nitrogen content, iodide value, loss on drying, pH, sulphated ash and available iodine as per BP 2019 are performed in well-equipped lab of BRiCM to review the test results with the acceptance criteria stated in the specification.
* Impurity testing of PVP-I as 1-Vinyl-2-pyrrolidinone, 2-Pyrrolidinone according to British Pharmacopeia (BP) 2019 and heavy metal (Pb) as per AOAC is carried out using HPLC, LC-MS-MS, AAS & ICPMS.
* Sterile water, the diluent of 0.6% PVP-I solution is characterized by performing the tests of pH, conductivity, total organic carbon, heavy metal (Pb, As) as per AWWA, endotoxin as per EU 85 and microbial count as per AOAC in the well-equipped Microbiology Lab of BRiCM.
* Production of 0.6% PVP-I Oro-nasal spray solution from batch dispensing to final product packing is carried out following the norms of cGMP
* In-process quality assurance/control of the product is done at real time by performing, volume check, pH of the solution, available iodine, UV absorbance as per BP 2019 and packing integrity with necessary primary and secondary packing materials.

Stability Study & Shelf-life estimation

* Stability studies of the product are carried out at both accelerated condition as well as real time condition as per ICH guidelines applicable for Stability Zone IVa.
* Stability studies at accelerated condition is carried out at 40 deg. C up to 12 months in 2 months interval and stability studies at real time condition is carried out at 25 deg. C up to two years in three months interval.
* Stability indicting parameters such as appearance, pH, available iodine, UV absorbance are included in both stability studies.
* Findings of both accelerated and real time stability studies are used to predict the shelf-life of the product up to two years.

Period of study The study will be carried out during the period of May 2020 to June 2021. Place of study Dhaka Medical College Hospital, Kurmitola General Hospital and Kuwait Moytree Hospital including product development & quality assurance will be held at Bangladesh Reference Institute for Chemical Measurements (BRiCM) Sampling Technique: Random sampling procedure will be followed using table of random numbers admitted patients of dedicated Covid-19 hospital like KGH, KMH and DMCH will be taken after fulfilling of inclusion and exclusion criteria. Then from interested participants written informed consent will be taken. After ward randomization will be carried out to select intervention group and control group.

Sampling Unit: Individual study subject i.e. selected each participants will be considered as a sample unit.

Data Collection instrument and Technique : After receiving written permission from respective hospital authority face to face interview will also be taken. Study personnel at the site will enter data from source documents corresponding to a subject's visit into the protocol-specific paper CRF (Case report form). All data collected during the course of this study must be reviewed and verified for completeness and accuracy by the Investigator.

Availability and Retention of Investigation Records: The Investigator must provide interim study report with data at every three months interval to the principle investigator. As per requirement study report and data may be provided to BMRC and DGDA. The Investigator must ensure the reliability and availability of source documents from which the information on the CRF will be derived. All study documents (patient files, signed informed consent forms, copies of CRFs, Study File Notebook, etc.) must be kept secured for a period of five years.

Data safety & Monitoring: Monitoring visits will be conducted by principle investigator, co- investigator as well as the representatives according to Guidelines for GCP. By signing this protocol, the investigator grants permission to the appropriate regulatory authorities to conduct on-site monitoring and/or auditing of all appropriate study documentation.

Subject Confidentiality:In order to maintain subject confidentiality, only a site number, subject number and subject initials will identify all study subjects on CRFs and other documentation submitted to the investigator. Additional subject confidentiality issues (if applicable) are covered in the Clinical Study Agreement.

Risk Management Plan: Bangasafe (proposed name) oro-nasal spray containing comparatively very low concentration (0.6% of PVP-I) is supposed to be safe in oro-nasal application. Moreover, this oro-nasal spray is intended to be used in the selected hospitalized patients under the direct supervision of doctors & nurses. Therefore, any adverse reaction risk if arises will be managed accordingly with the available facilities in respective hospital without any cost.

* If any discomfort, irritation, burning sensation occur then nasal irrigation with sterile plan water by 50 cc disposable syringe is to be given.
* If any hypersensitivity reaction occurs then anti-histamine and/or steroid is to be given

Clinical Laboratory Measurements Blood Chemistry Profile Blood sample for Group - C participants will be collected and sent to the respective hospitals/BRICM clinical chemistry lab for determining of TSH, FT3, FT4, Serum creatinine, alanine aminotransferase (ALT/SGPT) level including urine test.

Utilization of Results:By providing information and assurance about the efficacy and safety of 0.6% PVP-I , we can inform and encourage people to use it as oronasal spray safely for prevention of COVID-19, as an adjunct to PPE and reduce transmissibility of SARS Cov-2 virus.

ELIGIBILITY:
A. Moderately ill COVID-19 patient and asymptomatic to mild COVID-19 patent having multiple comorbidity

Inclusion Criteria

1. Hospital admitted patients tested positive COVID-19 within 24 hours in the laboratory by RT-PCR.
2. Patients with asymptomatic, mild to moderate illness of COVID-19.
3. Age group 18 year and above.
4. Consent of the patients, wish to be included in the study willingly.

Exclusion Criteria:

1. Patients with critical COVID-19 and moderate COVID-19 with other complication.
2. Patients having thyroid dysfunction, pregnant or lactating mother.
3. It should not be used prior to or after radioiodine scintigraphy or radioiodine treatment of thyroid carcinoma.
4. Patients allergic to iodine should be avoided
5. Have participated in other clinical study
6. Subjects with other severe acute or chronic conditions that may increase the risk of participation in the study and study treatment, or may interfere with interpretation of study results, and judged by the investigator as not suitable for participation in this clinical trial.

B. Healthy Individual

Inclusion Criteria:

1. Healthy individual (non COVID-19)
2. Age -18 years and above (as below18 years lesser concentration of drug may be required).
3. Consent of the participants who wish to participate.

Exclusion criteria:

1. Participants who has any major comorbidity.
2. Participants having thyroid dysfunction, pregnant or lactating mother.
3. It should not be used prior to or after radioiodine scintigraphy or radioiodine treatment of thyroid carcinoma.
4. Participants allergic to iodine should be avoided
5. Have participated in other clinical study
6. Subjects with other severe acute or chronic conditions that may increase the risk of participation in the study and study treatment, or may interfere with interpretation of study results, and judged by the investigator as not suitable for participation in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 798 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Viral concentration assessment in Naso-Oropharynx by applying 0.6% PVP-I on COVID-19 positive, moderately ill admitted patient | 24 hours
  Application of 0.6% PVP-I spray once (2 puff 0.6% PVP-I in each nostril and 2 puff inside mouth) to experimental group and distilled water to control group. Then follow up (waiting for 2-5 minutes) and collection of nasopharyngeal and oropharyngeal sawab for RT-PCR test for both group to assess viral concentration. Observation of the patients for 30 minutes for possible early adverse effects (if any) and subsequent management (if needed).
Effectiveness of 0.6% PVP-I assessment through viral concentration measurement | 24 hours
  Selection of 20 patients randomly with no or mild symptoms and obtain their consent for the further tests. Then application of 0.6% PVP-I spray 4 times (2 puff 0.6% PVP-I containing oronasal spray to each nostril and 2 puff inside mouth). Then collection of 2nd, 3rd and 4th sample from nasopharynx and oropharynx hourly for RT-PCR test to assess the viral concentration.

SECONDARY OUTCOMES:
TSH, FT3, FT4 and Unirine iodine concentration determination for assessing side effect on thyroid function after using 0.6% PVP-I oronasal spray on healthy volunteer | 10 Days
  Selection of 10 healthy volunteers randomly who will be selected for using 0.6% PVP-I Oro-Nasal spray 2 puff inside both nostrils and mouth 3 to 4 times a day for one month. Then collection of blood & urine of participants on day 0, 10, 20, 30 for determination of any change in thyroid functions like TSH, FT3, FT4 and Unirine iodine
Serum creatinine concentration determination for assessing side effect on kidney function after using 0.6% PVP-I oronasal spray on healthy volunteer | 10 Days
  Selection of 10 healthy volunteers randomly who will be selected for using 0.6% PVP-I Oro-Nasal spray 2 puff inside both nostrils and mouth 3 to 4 times a day for one month. Then collection of blood & urine of participants on day 0, 10, 20, 30 for determination of any change in kidney and liver functions Serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Kamal Arefin, Dr., Principal Investigator — Indoor Medical Officer, Department of ENT & Head-Neck Surgery, Dhaka Medical College Hospital
Locations (4):
- Bangladesh (4):
  - Bangladesh Reference Institute for Chemical Measurements, Dhaka, Dhanmondi
  - Dhaka Medical College Hospital, Dhaka
  - Kurmitola General Hospital, Dhaka
  - Kuwait-Moitree Hospital, Dhaka

IPD SHARING:
Plan to Share IPD: Yes
After completion of the project, a manuscript will be prepared and will be shared to the journal authority for publication. Data will be shared with the journal authority and make public as part of the publication.
Supporting Information: SAP, ICF, CSR
Time Frame: 3 months
Access Criteria: Available on public domain like figure share, research gate, Linkdin and others

DOCUMENTS (3):
  • Study Protocol (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT04872686/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT04872686/SAP_001.pdf
  • Informed Consent Form (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT04872686/ICF_002.pdf